CLINICAL TRIAL: NCT05192278
Title: Comparison of Different Volumes Spread of Erector Spinae Block in Post Mastectomy Pain Syndrome Management: A Randomized Controlled Trial
Brief Title: Comparison of Different Volumes Spread of Erector Spinae Block in Post Mastectomy Pain Syndrome Management
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, assist. prof. of anesthesia and pain management, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.21.11.1523
Record Dates: First submitted 2021-12-13; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 20 ml (Active Comparator): receive ESB with 1mL of methylprednisolone 40mg/mL with 10 mL of 0.5% bupivacaine and 2mL of nonionic contrast in 7 ml saline 0.9% (total 20 ml with bupivacaine 0.25%).
  Interventions: Other: erector spinae block
- Group 30 ml (Active Comparator): receive ESB with 1mL of methylprednisolone 40mg/mL with 15 mL of 0.5% bupivacaine and 2mL of nonionic contrast in 12 ml saline 0.9% (total 30 ml with bupivacaine 0.25%).
  Interventions: Other: erector spinae block

INTERVENTIONS:
Other: erector spinae block — The patients will do the procedure under fluoroscopic guidance. The patients were placed in prone position. After the identification of the T4 transverse process, the targeted injection site was anesthetized with 3-4 ml of 2% lidocaine. A 25-gauge spinal needle was advanced until it contacted the transverse process at the T4 level. Next, a solution of 1mL of methylprednisolone 40mg/mL with 7 mL of 0.25% bupivacaine and 2mL of nonionic contrast in 10 ml saline 0.9% (group A) and in 20 ml saline 0.9% (group B) will injected. Then another photo will be taken with the fluoroscopy to determine the level of spread in each group. After finished, the patients will transfer to the post-operative care unit and will monitored for any complication for one hour.

SUMMARY:
Cancer breast is one of the most common tumors among women and surgery is still the key for its management and cure. Post-mastectomy pain control is crucial as acute postoperative pain is a significant factor in the development of persistent chronic pain in the form of post-mastectomy pain syndrome.

Post-mastectomy pain syndrome (PMPS) is a common complication after breast cancer surgery and is often challenging to manage. It is estimated that PMPS occurs in 20%-44% of patients after breast surgery.

Adequate pain control for PMPS has become one of the most important goals and recently can achieve by multiple tools including multimodal analgesia and regional techniques.

Erector spinae block (ESB) is one of the new described regional techniques. Although its mechanism is not clear, the published data agree that it is promising block for chronic and acute pain and its simplicity and safety compared with thoracic epidural or bilateral paravertebral blocks.

ESB can be performed using a superficial approach between the large rhomboid muscle and the erector spinae muscle or the deep method beneath the erector spinae.

The use of the ESPB for chronic pain has recently expanded for various neuropathic pain conditions. Also, it reported with several volumes range from 10 to 30 ml of total volume.

DETAILED DESCRIPTION:
This prospective randomized open comparative study will be conducted in pain clinic, Mansoura University Hospitals. The study will be approved by the Ethics Research Committee of the Faculty of Medicine, Mansoura University and will be carried out in compliance with the Helsinki Declaration. Informed written consent will be signed from every patient participating in this study after full description of all details of every aspect in this study.

Patients more than 18 years old of both genders with PMPS not responding to medical treatments, and numeric rating scale (NRS) ≥ 4 that ranged from 0 (no pain) to 10 (extreme pain)., American society of Anesthesiology Physical Status class I and II, and Body mass index ˂ 30 were included in this study.

The exclusion criteria are patient refusal, local or systemic sepsis, coagulopathy, unstable cardiovascular and respiratory diseases, previous neurological deficits, history of psychiatric disorders, history of drug abuse, distorted local anatomy, and those who were allergic to the used medications were excluded from the study.

All the patients will inform about the numerical rating score (NRS) from zero to 10 (where 0 no pain, 10 the worst pain) to describe their pain.

Random selection of patients:

The study participants were randomly grouped on a scale of 1:1, using a computer-generated list of random numbers. The distribution results were sealed in an opaque envelope and kept by the study administrator. On the day of block, the study manager handed the envelope to the anesthesiologist who will perform the block.

Grouping:

Group A: receive ESR with 1mL of methylprednisolone 40mg/mL with 10 mL of 0.5% bupivacaine and 2mL of nonionic contrast in 7 ml saline 0.9% (total 20 ml with bupivacaine 0.25%).

Group B: receive ESR with 1mL of methylprednisolone 40mg/mL with 15 mL of 0.5% bupivacaine and 2mL of nonionic contrast in 12 ml saline 0.9% (total 30 ml with bupivacaine 0.25%).

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years old of both genders
* with post-mastectomy pain syndrome not responding to medical treatments,
* and numeric rating scale (NRS) ≥ 4 that ranged from 0 (no pain) to 10 (extreme pain).,
* American society of Anesthesiology Physical Status class I and II,
* and Body mass index ˂ 30 were included in this study

Exclusion Criteria:

* patient refusal,
* local or systemic sepsis,
* coagulopathy,
* unstable cardiovascular
* and respiratory diseases,
* previous neurological deficits,
* history of psychiatric disorders,
* history of drug abuse,
* distorted local anatomy,
* and those who were allergic to the used medications

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
The level spread of each volume. | immediately after injection. C arm photo will be taken to know the level of distribution
  The level spread of each volume.
Numerical analogue scale | after 4 weeks from procedure
  from 0 (no pain) to 10 (sever pain)
Numerical analogue scale | after 8 weeks from procedure
  from 0 (no pain) to 10 (sever pain)
Numerical analogue scale | after 12 weeks from procedure
  from 0 (no pain) to 10 (sever pain)

SECONDARY OUTCOMES:
Patient satisfaction | after 4 weeks from the procedure
  evaluated by using a linear scale in which 0 is very dissatisfied and 10 is very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Nevert adel, Al Mansurah, Egypt

REFERENCES:
- [Derived] Abdelghaffar NA, Amer GF. Comparison of different volumes spread of erector spinae block in postmastectomy pain syndrome management: a prospective randomized comparative study. BMC Anesthesiol. 2023 Aug 22;23(1):282. doi: 10.1186/s12871-023-02239-1. PMID 37608269